CLINICAL TRIAL: NCT00145990
Title: The Impact of Dosimeter on Measurement of Airway Responsiveness to Methacholine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 257-2005
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: methacholine PC20; dosimeter; asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

INTERVENTIONS:
Drug: methacholine
Device: KoKo Digidoser
Device: Rosethal Dosimeter

SUMMARY:
To determine whether there is a difference in two different breathing tests used to detect asthma. Hypothesis: The Digidoser delivers less methacholine to the airways and will result in a higher PC20 than the value determined by the Rosenthal Dosimeter.

DETAILED DESCRIPTION:
Bronchoprovocation with methacholine is used to confirm the diagnosis of asthma. The procedure involves inhaling methacholine through a nebulizer attached to a dosimeter that delivers a precise volume of methacholine. The endpoint of the test is the provocational concentration that produces a 20% decrease in FEV1 (PC20). To standardize the procedure, the American Thoracic Society (ATS) recommends that the nebulizer output be calibrated to deliver an output of 0.9 ± 0.09 mL/min.

The Rosenthal Dosimeter and the KoKo Digidoser are two commonly used dosimeters. In an attempt to follow the ATS guideline we discovered that the nebulizer output was lower with the KoKo Digidoser and could not be calibrated. However, it is unclear whether the apparent lower output is a result of the Digidoser delivering less solution or that the ATS method of determining output is not applicable to this dosimeter. To answer this question, we propose to determine the methacholine PC20 in subjects with asthma using the two dosimeters. It is our hypothesis that the Digidoser delivers less methacholine and thus will produce a higher PC20 than the Rosenthal Dosimeter.

Twelve nonsmoking subjects with mild asthma will be selected on the basis of > 18 years of age, a baseline FEV1 of > 60% predicted and a screening PC20 of < 8mg/ml. Subjects will be randomized to perform a methacholine challenge with the Digidoser and the Rosenthal Dosimeter on two different days in an unblinded, crossover manner. The geometric mean PC20 with each dosimeter will be compared with a paired t test. The results of this study will indicate whether the Digidoser has the potential of causing false negative test results or whether the ATS method of determining output should not be used with this dosimeter.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female >18 years of age, with a previous diagnosis of asthma.
* Women of child bearing age must not be pregnant or nursing and be using an acceptable method of contraception.
* Screening FEV1 > 70% of predicted for height, age, sex, and race when bronchodilators are withheld for appropriate intervals.
* At least a 20% decrease in FEV1 after inhaling ≤ 8 mg/ml of methacholine (i.e., a PC20 FEV1 ≤8 mg/ml) using the KoKo Digidoser system.
* Ability to perform ATS-acceptable and reproducible spirometry.

Exclusion Criteria:

* Cigarette smoking in past year or > 10 pack year smoking history.
* Respiratory tract infection within the last four weeks.
* History of severe asthma attack requiring hospitalization in the previous 12 months.
* Short course of oral corticosteroids in the past 3 weeks.
* Inability to withhold caffeinated beverages for 12 hours or medications for appropriate intervals prior to each methacholine challenge.
* If female, a positive urine β-HCG test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Geometric mean PC20 methacholine for each dosimeter method.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen Khan, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States